CLINICAL TRIAL: NCT06687577
Title: Dialectical Behavior Therapy for Smoking Cessation in High Risk Veterans
Brief Title: DBT for Smoking Cessation in High Risk Veterans
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Veterans Medical Research Foundation (Other)
Collaborators: University of California (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 101760002
Record Dates: First submitted 2024-01-24; First posted 2024-11-13 (Actual); Last update posted 2026-01-08 (Actual); Status verified 2025-09

CONDITIONS: Tobacco Dependence; Suicidal
MeSH Terms: conditions — Tobacco Use Disorder | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: Participants are randomized to DBT or to treatment as usual (TAU)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- DBT (Experimental): Standard behavioral cessation intervention adapted to incorporate DBT skills for emotion regulation.
  Interventions: Behavioral: DBT-C
- TAU (Active Comparator): Standard behavioral cessation intervention.
  Interventions: Behavioral: Treatment as usual

INTERVENTIONS:
Behavioral: DBT-C — Tobacco cessation treatment adapted for high risk population.
  Arms: DBT
Behavioral: Treatment as usual — Standard behavioral tobacco cessation treatment.
  Other Names: TAU
  Arms: TAU

SUMMARY:
Individuals prone to suicidality are typically excluded from tobacco cessation interventions even though they are disproportionately likely to smoke, and even though smoking cessation has been linked to improved mood and reduced risk of suicide.

This trial enrolls Veteran smokers at high risk for suicide, and assigns them to receive either cessation treatment as usual, or a novel treatment that incorporates standard behavioral cessation treatment with Dialectical Behavior Therapy (DBT), an evidence-based treatment for suicide risk.

DETAILED DESCRIPTION:
Individuals with behavioral health problems are a significant tobacco-related health disparity group in that they are more likely to use tobacco and evidence disproportionate consequences from their use. Cigarette smoking or usage of other nicotine products is strongly associated with symptoms of emotional distress, while cessation is associated with significant reductions in symptoms of anxiety and depression and improved mental health functioning. Individuals with who have difficulty managing negative emotions (emotional dysregulation) may be especially vulnerable to tobacco dependence and have particular difficulties with smoking cessation. Because cessation studies commonly exclude smokers exhibiting emotional dysregulation (such as recent suicidality and/or acute emotional instability), little extant evidence is available to inform optimal treatment approaches for these smokers.

Dialectical behavior therapy skills group (DBT-SG) is an evidence-based approach to addressing dysregulation of emotion, teaching skills to help manage emotions more effectively. Preliminary empirical work suggests DBT may also be an effective approach to addressing smoking cessation. Difficulty managing negative emotions is a common reason for smoking cessation failure, suggesting that group DBT may be an effective intervention for cessation. Investigators propose to conduct a pilot treatment study with veterans at risk for suicide as an initial step to developing and evaluating the utility of DBT for smoking cessation in subgroups with high levels of emotion dysregulation.

The primary aims of the proposed study are to 1) adapt a 12-week, manualized DBT-based group intervention for smoking cessation (DBT-C); 2) conduct a randomized trial testing whether DBT-C has better smoking cessation outcomes than standard smoking cessation treatment (SCCT); 3) evaluate whether DBT-C participants have greater improvements on measures of emotion regulation, mood and suicidality than those in the SSCT conditions; and 4) examine intervention acceptability and feasibility.

ELIGIBILITY:
Inclusion Criteria:

* Veteran receiving VA healthcare
* multiple indicators of elevated suicide risk in 6 month period

Exclusion Criteria:

* cognitive impairment
* unable to attend virtual intervention

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 67 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Proportion of participants who stop using tobacco | 6 months
  Reduction in use or abstinence

SECONDARY OUTCOMES:
Average change per participant in quality of sleep | 6 months
  Change in sleep quality/quantity will be evaluated using the Insomnia Severity Index (ISI), a brief, valid measure of sleep quality. The ISI will be administered at baseline, end of treatment, and end of follow-up.
  Morin et al. (2011). The Insomnia Severity Index: psychometric indicators to detect insomnia cases and evaluate treatment response. Sleep 34(5), 601-8.
Average improvement in physical pain per participant | 6 months
  Participants will self-report frequency of pain on scale from 0 (rarely/never) to 7 (always/almost always). They will self-report pain intensity on a similar scale from 0 (no/mild pain) to 7 (severe pain). These measures are completed at baseline, end of treatment, and end of follow-up.
Average improvement in negative mood per participant | 6 months
  Change in negative mood will be evaluated via the Positive and Negative Affect Schedule (PANAS), administered at each assessment point. The PANAS asks respondents to indicate the extent to which a series of 10 positive and 10 negative affect terms have applied to them over the past 2 weeks.
  Watson et al (1988). Development and validation of brief measures of positive and negative affect: The PANAS scales. J Pers Soc Psychol, 54(6), 1063.

CONTACTS AND LOCATIONS:
Overall Officials: Neal M. Doran, Principal Investigator — Veterans Medical Research Foundation / VA
Locations (1):
- Veterans Medical Research Foundation, San Diego, California, United States

IPD SHARING:
Plan to Share IPD: No
Anonymized data may be made available upon request from the PI if approved by the sponsor.